CLINICAL TRIAL: NCT02090101
Title: Phase II Study Evaluating the Influence of LV5FU2 Bevacizumab Plus Anakinra Association on Vascularization of Liver Metastases of Metastatic Colorectal Cancer: Proof of Concept Study
Brief Title: Study Evaluating the Influence of LV5FU2 Bevacizumab Plus Anakinra Association on Metastatic Colorectal Cancer
Acronym: IRAFU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-003367-55
Record Dates: First submitted 2014-03-13; First posted 2014-03-18 (Estimated); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ANAKINRA (Experimental): LV5FU2 + bevacizumab + anakinra
  Interventions: Drug: ANAKINRA

INTERVENTIONS:
Drug: ANAKINRA

SUMMARY:
The metastatic colon cancer is a major public health problem despite advances in chemotherapy; few new drugs are in development for the treatment of this pathology.

Many studies have shown that human colon cancer is a tumor that is recognized by the immune system and the presence of lymphocytic infiltrates in the tumor bed is associated with a better prognosis. Conversely, the effect of chemotherapy on the immune response is little studied.

Recently the importance of myeloid suppressor cells (MDSC) in the development of colon cancer and the effect of 5- fluorouracil on this cell population has been highlighted. An accumulation of these cells in the blood and lymphoid organs during tumor progression is observed. Moreover, it has been established that the death of MDSC induced by 5-fluorouracil induces activation of caspase -1 and IL-1beta by these MDSC.

These events promote the polarization of CD4 T cells in intratumoral Th17 lymphocytes. The IL- 17 produced by these cells exerts a pro-angiogenic effect in inducing proliferation of endothelial cells expressing and thus limits the effect of 5- fluorouracil endoglin.

In humans, it has also been observed that chemotherapy using 5- fluorouracil and in particular LV5FU2 association +/- bevacizumab induces rapid death of blood MDSC as well as activation of caspase 1 in these cells. Thus, production of IL - 1 is detected in the serum of patients after 24 hours of the administration of 5-fluorouracil.

Chronic inflammation and the production of interleukin- 1 can alter the effectiveness of anti -tumor immune responses and facilitate angiogenesis. Many preclinical data suggest a role of anti -tumor inhibition of IL- 1beta, but the effect of a combination of chemotherapy and an inhibitor of IL - 1beta has not yet been tested in human.

Anakinra is a drug used in humans for many years to treat signs and symptoms of rheumatoid arthritis. In combination with methotrexate, in patients whose response to methotrexate alone is not satisfactory it had shown interesting results. The dose used clinically is 100 mg per day which is the dose that is proposed to be tested in this study.

In this context it should be remembered that methotrexate is a chemotherapeutic agent from the class of antimetabolites such as 5- fluorouracil.

RCP of this drug indicate that in studies originator toxicity was similar between the control arm and anakinra arm with an increase in serious infections (1.8 % vs 0.7 %) and an increased incidence of neutropenia (2.5 % neutropenia > grade = 1). The main toxicity observed is a painful inflammatory reaction at the injection site in 70 % of patients The investigators believe that this project could permit to validate in man preclinical observations showing an anti-tumor potential for combination anakinra and 5 fluorouracil.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Age ≥ 18 and ≤ 80 years
* Performance status of 0 or 1 according to the ECOG score of WHO
* Patient with Metastatic colorectal non-curative and progression on therapy in first -line therapy containing 5-fluorouracil and bevacizumab cancer.
* Patient with low or intermediate risk defined by modified Kohne's criteria
* Hepatic metastases ≥ 1 cm
* Evaluation Review (CT chest, abdomen and pelvis ) made in the previous 4 weeks and showing the presence of a measurable lesion according to RECIST 1.1 criteria.
* Indication treatment LV5FU2 + bevacizumab validated
* Patient whose understanding of the study is good
* Biological values within the following limits :

  * Bilirubin ≤ 1.5 x upper limit of normal ( N)
  * AST and ALT ≤ 5 N
  * Creatinin ≤ 1.5 N and creatinin clearance > 60 ml / min
  * Neutrophils ≥ 1.5 . 109 / L
  * Platelets ≥ 100 . 109 / L
  * Hemoglobin ≥ 9 g / dL ( even if includable patients were transfused ) .
  * Albumin ≥ 30 g / L
  * Serological hepatitis B , C and HIV negative
* Information given and signed informed consent
* Patient affiliated to a social security system
* For women of childbearing age , the need for effective contraception.

Exclusion Criteria:

Related to the disease:

* Other cancer within 5 years prior to entry into the trial or concomitant (except carcinoma in situ of the cervix or basal cell carcinoma of the skin ) .
* Presence of brain metastasis
* Prognosis estimated survival <3 months

Related to treatment :

* Presence of a contraindication to bevacizumab ( major surgery in the previous 28 days , the risk of arterial thrombosis, risk of bleeding , deep vein thrombosis without effective anti- coagulant treatment or unbalanced anticoagulant treatment) Concomitant systemic
* Immunotherapy , immunosuppressants, corticosteroids ≥ 1mg/kg or hormone therapy : corticosteroids administered chronically , immunosuppressive therapy, biotherapy administered under the management of inflammatory disease (anti -TNF , anti- IL6 ... )
* Hypersensitivity to one of the compounds of treatments
* Latex Hypersensitivity ( the cap of the syringe containing anakinra contains dry natural rubber, a derivative of latex), which may cause allergic reactions
* Peripheral neuropathy grade ≥ 2
* History of autoimmune disease or inflammatory

Related to patient conditions :

* Participation during or within 30 days prior to study entry to another clinical trial with an experimental molecule.
* Serious disease unbalanced, underlying infection that may prevent the patient from receiving treatment
* Intestinal occlusion or sub- occlusion or history of inflammatory bowel disease
* Pregnancy (test mandatory inclusion pregnancy) , lactation or lack of effective contraception for men and women of childbearing age
* Psychiatric disease compromising understanding of the information or the accomplishment of the study
* Patient under guardianship, curatorship or judicial protection
* Unable to sign the informed consent or to submit to medical follow-up for geographical, social or psychological reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-10-10 (Actual); Primary Completion 2014-10-10 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Response rate after 2 months in patients with colorectal cancer with liver metastases treated with anakinra and LV5FU2/bevacizumab | after 2 months of treatment

SECONDARY OUTCOMES:
Response rate by echography | 15 days after the beggining of treatment
Tumor control rate | At 2, 4, 6, 9 and 12 months after the beginning of treatment
Overall survival | At 2, 4, 6, 9 and 12 months after the beginning of treatment
Rate and safety profile according to NCI-CTCAE v4 | Every 15 days before each cycle of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges François Leclerc, Dijon, Burgundy, France